CLINICAL TRIAL: NCT02626000
Title: A Phase 1b/3 Multicenter, Randomized, Trial of Talimogene Laherparepvec in Combination With Pembrolizumab for the Treatment of Subjects With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Talimogene Laherparepvec With Pembrolizumab for Recurrent Metastatic Squamous Cell Carcinoma of the Head and Neck (MASTERKEY232 / KEYNOTE-137)
Acronym: MASTERKEY232
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130232; 20130232 / KEYNOTE-137 (Other: Merck / Amgen); 2015-003011-38 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-12-10 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma of the Head and Neck
Keywords: Recurrent Metastatic Squamous Cell Carcinoma Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — talimogene laherparepvec; pembrolizumab

STUDY DESIGN:
Masking Description: For Phase 1b there are no 'maskings' as it's open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talimogene Laherparepvec + Pembrolizumab (Experimental): Talimogene laherparepvec is administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL on day 1 followed by a dose of 10⁸ PFU/mL 3 weeks after the initial dose and every 3 weeks (Q3W) thereafter. Pembrolizumab is administered by intravenous infusion at a dose of 200 mg Q3W after the initial dose. Participants are treated until complete response, no injectable lesions, confirmed disease progression, intolerance of study treatment, 24 months from the date of the first dose of talimogene laherparepvec, or end of study, whichever occurred first.
  Interventions: Drug: Talimogene Laherparepvec; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Talimogene Laherparepvec — The initial dose of talimogene laherparepvec is up to 8.0 mL of 10⁶ PFU/mL. Subsequent doses of talimogene laherparepvec are up to 8.0 mL of 10⁸ PFU/mL.
  Other Names: IMLYGIC®
Biological: Pembrolizumab — Administered as a 30-minute intravenous infusion at a dose of 200 mg Q3W
  Other Names: KEYTRUDA®

SUMMARY:
The primary objective of this study was to evaluate the safety, as assessed by incidence of dose limiting toxicity (DLT), of talimogene laherparepvec in combination with pembrolizumab in adults with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
This is a phase 1b/3, multicenter, clinical trial conducted in 2 parts (phase 1b and phase 3). In phase 1b talimogene laherparepvec is to be administered in combination with pembrolizumab to adults with recurrent or metastatic squamous cell carcinoma of head and neck (SCCHN). Dose limiting toxicity (DLT) is to be evaluated based on the first 18 DLT-evaluable participants. An expansion cohort of up to an additional 22 treated patients could be enrolled to further evaluate the safety and to estimate the efficacy of the combination of talimogene laherparepvec with pembrolizumab and to support a decision to initiate the phase 3 part of the study. The phase 3 part of the study was designed as a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, as assessed by overall survival, of treatment with talimogene laherparepvec with pembrolizumab versus placebo with pembrolizumab in adults with recurrent or metastatic SCCHN, however, a decision was made not to proceed to the phase 3 part of the study.

ELIGIBILITY:
Inclusion Criteria

* Male or female age ≥ 18 years at the time of informed consent
* Histologically confirmed diagnosis of metastatic or recurrent SCCHN of the oral cavity, oropharynx, hypopharynx, or larynx. Disease must be unsuitable for curative surgical resection and must not be amenable to curative radiotherapy.
* Disease must have progressed after treatment with a platinum-containing regimen and should be defined as one of the following:

  i. disease progression or recurrence between 3 to 6 months of prior curatively intended multimodal therapy (which includes platinum therapy) for locoregionally advanced SCCHN.

ii. disease progression or recurrence after prior platinum therapy in the recurrent or metastatic setting Note: This criterion is only applicable for subjects who have not had treatment in the recurrent/metastatic setting

* Subject must be candidate for intralesional therapy administration defined as one or more of the following:

  i. at least 1 injectable cutaneous, subcutaneous, or nodal SCCHN tumor ≥ 10 mm in longest diameter ii. multiple injectable cutaneous, subcutaneous, or nodal SCCHN tumors that in aggregate have a longest diameter of ≥ 10 mm Note: Mucosal surfaces of tumor lesions and visceral metastases should not be injected.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function determined within 14 days prior to enrollment
* Female subject of childbearing potential must have a negative pregnancy test within 72 hours prior to enrollment.
* Other Inclusion Criteria May Apply

Exclusion Criteria

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Primary nasopharyngeal carcinoma.
* Subject at risk of airway compromise in the event of postinjection tumor swelling/inflammation based on investigator judgment.
* Phase 3: Previous treatment with 3 or more systemic regimens given for recurrent and/or metastatic disease
* History of other malignancy within the past 3 years
* History of interstitial lung disease (ILD).
* Prior therapy with talimogene laherparepvec, pembrolizumab, other anti-PD-1, any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathway.
* History or evidence of active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Evidence of clinically significant immunosuppression
* Active herpetic skin lesions or prior complications of herpetic infection (eg, herpetic keratitis or encephalitis).
* Requires intermittent or chronic treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.
* Prior chemotherapy, radiotherapy, biological cancer therapy, targeted therapy, or major surgery within 28 days prior to enrollment or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
* Expected to require other cancer therapy while on study with the exception of local palliative radiation treatment to the site of bone and other metastasis.
* Known human immunodeficiency virus (HIV) disease.
* Has acute or chronic active hepatitis B virus or hepatitis C virus infection or received treatment with nucleotide analogs such as those used in the treatment of hepatitis B virus (eg, lamivudine, adefovir, tenofovir, telbivudine, entecavir), ribavirin, or interferon alpha within 12 weeks of initiation of study treatment.
* Received live vaccine within 28 days prior to enrollment.
* Subject is pregnant or breast-feeding, or expecting to conceive or father children within the duration of the trial
* Female subject of childbearing potential or male subject of reproductive potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec/placebo or 4 months after the last dose of pembrolizumab, whichever is later.
* Sexually active subjects or their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec/placebo.
* Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for herpes simplex virus type 1 (HSV-1)-induced complications (eg, immunosuppressed individuals, HIV-positive individuals, pregnant women, or children under the age of 1 year) during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec
* Has history of (non-infectious) pneumonitis that required steriods or current pneumonitis
* Subjects with tumor that directly contacts or encases a major blood vessel AND there is ulceration and/or fungation onto the skin surface
* History of re-irradiation to a field which includes the carotid arteries
* Other Exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (29):
- United States (6):
  - Research Site, Newark, Delaware
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Billings, Montana
  - Research Site, New York, New York
  - Research Site, Canton, Ohio
- Australia (2):
  - Research Site, Geelong, Victoria
  - Research Site, Melbourne, Victoria
- Research Site, Salzburg, Austria
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Wilrijk
- Research Site, Toronto, Ontario, Canada
- France (3):
  - Research Site, Bordeaux
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
- Greece (2):
  - Research Site, Athens
  - Research Site, Ioannina
- Research Site, Milan, Italy
- Spain (3):
  - Research Site, Seville, Andalusia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Madrid
- Switzerland (3):
  - Research Site, Bellinzona
  - Research Site, Geneva
  - Research Site, Zurich
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Oxford
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Harrington KJ, Kong A, Mach N, Chesney JA, Fernandez BC, Rischin D, Cohen EEW, Radcliffe HS, Gumuscu B, Cheng J, Snyder W, Siu LL. Talimogene Laherparepvec and Pembrolizumab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (MASTERKEY-232): A Multicenter, Phase 1b Study. Clin Cancer Res. 2020 Oct 1;26(19):5153-5161. doi: 10.1158/1078-0432.CCR-20-1170. Epub 2020 Jul 15. PMID 32669371
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 centers in Australia, Canada, Europe, and the United States.
  This study was designed to be conducted in 2 parts (phase 1b and phase 3). A decision was made not to initiate the phase 3 part of the study.
Groups:
- Talimogene Laherparepvec + Pembrolizumab: Talimogene laherparepvec was administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL on day 1 followed by a dose of 10⁸ PFU/mL every 3 weeks (Q3W) thereafter. Pembrolizumab was administered by intravenous infusion at a dose of 200 mg Q3W.
  Participants were treated until complete response, no injectable lesions, confirmed disease progression, intolerance of study treatment, 24 months from the date of the first dose of talimogene laherparepvec, or end of study, whichever occurred first.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Started | 36
Completed | 6
Not Completed | 30
Not completed — Decision by Sponsor | 1
Not completed — Death | 29

BASELINE CHARACTERISTICS:
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 21
  ≥ 65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black (or African American) | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 33
  Other | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 9
    1 (Restricted but ambulatory) | 27
Herpes Simplex Virus Status [Count of Participants; unit: Participants]
  Negative | 5
  Positive | 22
  Unknown | 9
Primary Tumor Site [Count of Participants; unit: Participants]
  Oropharynx | 9
  Larynx | 4
  Oral Cavity | 20
  Hypopharynx | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: The following toxicities (graded per the Common Terminology Criteria for Adverse Events v 4.0) were considered DLTs if judged by the investigator to be related to either study drug:
  * grade 4 non-hematologic (non-laboratory) toxicity
  * ≥ grade 3 pneumonitis
  * grade 3 non-hematologic toxicity for > 3 days with optimal supportive care
  * grade 3 fatigue was not classified as DLT, regardless of duration
  * any ≥ grade 3 non-hematologic laboratory value if:
    * medical intervention was required,
    * the abnormality led to hospitalization, or
    * the abnormality persisted at ≥ grade 3 for > 1 week unless deemed not clinically important by investigator and sponsor
  * grade 3 or 4 febrile neutropenia
  * thrombocytopenia < 25 x 10⁹/L associated with bleeding event requiring intervention
  * serious herpetic event: herpetic encephalitis, encephalomyelitis, or disseminated herpetic infection
  * grade 5 toxicity
  * other intolerable toxicity leading to permanent discontinuation of either study drug.
Time Frame: First 6 weeks after the initial administration of talimogene laherparepvec and pembrolizumab in combination
Population: The DLT analysis set included DLT-evaluable participants who had the opportunity to be on treatment for at least 6 weeks and had received at least 2 doses of talimogene laherparepvec and 2 doses of pembrolizumab in combination, or who had a DLT during the DLT evaluation period after at least 1 dose of both study drugs in combination.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 16
Participants | 1

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a best overall response of complete response or partial response assessed by the investigator using immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Response was based on the size of tumors assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
  Complete response (iCR): Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response (iPR): Decrease in tumor burden ≥ 30% relative to baseline. Confirmation by a consecutive assessment at least 4 weeks after first documentation required.
  Analyses are presented below for both the unconfirmed and confirmed results.
Time Frame: Up to the primary analysis data cutoff date of 02 November 2017; median (minimum, maximum) time on follow-up was 14.36 (1.4, 67.0) weeks.
Population: The efficacy analysis set included all enrolled participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab, excluding participants with locoregionally advanced disease with a recurrence < 3 months after prior platinum-containing curatively intended multimodal therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
percentage of participants
  Confirmed Response | 9.4 [2.0 to 25.0]
  Unconfirmed Response | 15.6 [5.3 to 32.8]

3. Secondary Outcome: Complete Response Rate
Description: Complete response rate (iCRR) was defined as the percentage of participants with a best overall response of complete response assessed by the investigator using immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Response was based on the size of tumors assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
  Complete response (iCR): Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Analyses are presented below for both the unconfirmed and confirmed results.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
percentage of participants
  Confirmed Response | 0.0 [0.0 to 10.9]
  Unconfirmed Response | 0.0 [0.0 to 10.9]

4. Secondary Outcome: Best Overall Confirmed Response
Description: Best overall visit response of iCR, iPR, stable disease (iSD), progressive disease (iPD) or unevaluable (iUE) based on investigator assessment using irRECIST.
  iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new). Any pathological lymph nodes (target or non-target) must have reduction in short axis to <10 mm.
  iPR: Decrease in tumor size ≥ 30% relative to baseline. iPD: Increase in tumor size ≥ 20% and at least 5 mm absolute increase compared to nadir or qualitative worsening of non-target lesions or a new lesion.
  iSD: Neither sufficient shrinkage to qualify for iCR or iPR nor sufficient increase to qualify for iPD.
  iUE: Any baseline lesion which was not assessed or was unable to be evaluated leading to an inability to determine the status of that particular tumor.
  Not Done: Radiographic imaging was not performed to evaluate the response. iCR, iPR, and iPD required confirmation by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
Participants
  Complete Response (iCR) | 0
  Partial Response (iPR) | 3
  Stable Disease (iSD) | 10
  Progressive Disease (iPD) | 4
  Unevaluable (iUE) | 6
  Not Done | 9

5. Secondary Outcome: Duration of Confirmed Response
Description: Duration of response (iDOR) per irRECIST was defined as the time from the date of an initial response of iCR or iPR that was subsequently confirmed to the earlier of a participant overall response of iPD or death. Participants who did not end their response at the time of analysis were censored at their last evaluable tumor assessment.
Time Frame: as for outcome 2
Population: Enrolled participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab, excluding participants with locoregionally advanced disease with a recurrence < 3 months after prior platinum-containing curatively intended multimodal therapy, with a best response of iCR or iPR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 3
months | NA [NA to NA] — Could not be estimated due to the low number of events

6. Secondary Outcome: Disease Control Rate
Description: Disease control rate (iDCR) was defined as the percentage of participants with a best overall response of iCR or iPR or iSD assessed by the investigator using irRECIST.
  Complete response (iCR): Disappearance of all lesions (whether measurable or not and whether baseline or new) and confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial response (iPR): Decrease in tumor burden ≥ 30% relative to baseline. Confirmation by a consecutive assessment at least 4 weeks after first documentation required.
  Stable disease (iSD): Neither sufficient shrinkage to qualify for iCR or iPR nor sufficient increase to qualify for iPD.
  Analyses are presented below for both the unconfirmed and confirmed results.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
percentage of participants
  Confirmed Response | 40.6 [23.7 to 59.4]
  Unconfirmed Response | 40.6 [23.7 to 59.4]

7. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (iPFS) per irRECIST was defined as the interval from first dose to the earlier of a participant overall response of iPD or death from any cause; otherwise, iPFS was censored at the last evaluable tumor assessment. The initial date of an iPD that was consecutively confirmed was used.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
months | 3.0 [2.0 to 5.8]

8. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the interval from first dose to the event of death from any cause; otherwise, OS was censored at the date the participant was last known to be alive.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 32
months | 5.2 [2.1 to 11.4]

9. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of adverse events was assessed by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and based on the following scale:
  Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death.
  A serious adverse event is an AE that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From first dose of study drug to 30 days after last dose; the median (range) duration of treatment was 5.6 (0.1 to 75.3) weeks for talimogene laherparepvec and 6.1 (0.1, 105.3) weeks for pembrolizumab.
Population: All enrolled participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Talimogene Laherparepvec + Pembrolizumab: Talimogene laherparepvec (T-VEC) was administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL on day 1 followed by a dose of 10⁸ PFU/mL every 3 weeks (Q3W) thereafter. Pembrolizumab was administered by intravenous infusion at a dose of 200 mg Q3W.
  Participants were treated until complete response, no injectable lesions, confirmed disease progression, intolerance of study treatment, 24 months from the date of the first dose of talimogene laherparepvec, or end of study, whichever occurred first.
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
Number analyzed (Participants) | 36
Participants
  All treatment-emergent adverse events | 36
  Treatment-emergent adverse events grade ≥ 2 | 36
  Treatment-emergent adverse events grade ≥ 3 | 26
  Treatment-emergent adverse events grade ≥ 4 | 11
  Serious adverse events | 26
  AE leading to discontinuation of T-VEC | 6
  AE leading to discontinuation of pembrolizumab | 6
  Fatal adverse events | 7
  Talimogene laherparepvec-related AEs | 21
  Pembrolizumab-related AEs | 21

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose; the median (range) duration of treatment was 5.6 (0.1 to 75.3) weeks for talimogene laherparepvec and 6.1 (0.1, 105.3) weeks for pembrolizumab.
Description: Serious adverse event and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Talimogene Laherparepvec + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 29/36
Serious Adverse Events (participants affected / at risk) | 26/36
Other Adverse Events (participants affected / at risk) | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec + Pembrolizumab (N=36)
Dysphagia (Gastrointestinal disorders) | 2
Odynophagia (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
General physical health deterioration (General disorders) | 2
Mucosal haemorrhage (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection bacterial (Infections and infestations) | 1
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec + Pembrolizumab (N=36)
Anaemia (Blood and lymphatic system disorders) | 6
Ear pain (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Odynophagia (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 5
Face oedema (General disorders) | 2
Fatigue (General disorders) | 10
Influenza like illness (General disorders) | 5
Injection site pain (General disorders) | 3
Pyrexia (General disorders) | 12
Lower respiratory tract infection (Infections and infestations) | 4
Oral candidiasis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 3
Body temperature increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Headache (Nervous system disorders) | 6
Confusional state (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Weight decreased (Investigations) | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02626000/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02626000/SAP_002.pdf